CLINICAL TRIAL: NCT01828242
Title: The Empowerment Model Towards Type 2 Diabetic Adults To Enhance Vegetable Intake in Achieving Glycemic Control
Acronym: EDMID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SEAMEO Regional Centre for Food and Nutrition (Other)
Responsible Party: Principal Investigator, Tan Shot Yen, Medical Doctor, PhD Candidate (Nutrition), SEAMEO Regional Centre for Food and Nutrition
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Empowerment for DM
Record Dates: First submitted 2013-03-19; First posted 2013-04-10 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Glycemic Control for Diabetes Mellitus
Keywords: HbA1C

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Empowerment model to Diabetes (Experimental): Empowerment model to improve dietary intake
  Interventions: Behavioral: Empowerment model to improve dietary intake
- Control group following conventional approach (Active Comparator): Control group following conventional approach
  Interventions: Other: Control group following conventional approach

INTERVENTIONS:
Behavioral: Empowerment model to improve dietary intake — Empowerment model using specific guidelines to improve dietary intake
  Arms: Empowerment model to Diabetes
Other: Control group following conventional approach — Control group following conventional approach
  Arms: Control group following conventional approach

SUMMARY:
Life style changes, particularly in dietary patterns have contributed a great deal to the incidence and risks of type 2 Diabetes. Decreased intakes of vegetables and fruits replaced by pre processed food, added sugar and those of animal origin lead towards rapid increase of adult-onset-diabetes.

In spite of the knowledge of the benefit of consuming vegetable and fruits, and people are well informed, they still need to be committed to perform a behavior and implement these intention. Behavioral approach methods have demonstrated successful adherence in health education with life style changes.

Objective: To identify the impact of The Empowerment Model to enhance vegetable intake in Type 2 Diabetes Mellitus adults in achieving glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* fasting blood glucose ≥126 mg/dL
* HbA1C >8%

Exclusion Criteria:

* those who have serious, unstable medical conditions, or related to metabolic disorders (i.e. thyroid diseases)
* significant co-morbid illnesses such as liver disease, kidney disease, cancer, bowel diseases/ malfunction, pregnancy or nursing mothers.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
HbA1C | Baseline (week 0), Endline (week 12)

SECONDARY OUTCOMES:
Post Prandial blood glucose | Daily for 12 weeks
Fasting Blood Glucose | Daily for 12 weeks

OTHER OUTCOMES:
Iron status | Baseline (week 0), Endline (week 12)

CONTACTS AND LOCATIONS:
Overall Officials: Tan S Yen, MSc, Principal Investigator — SEAMEO-RECFON, University of Indonesia
Locations (1):
- Telecommunication Company, Jakarta, Jakarta Special Capital Region, Indonesia

REFERENCES:
- [Background] Yoon KH, Lee JH, Kim JW, Cho JH, Choi YH, Ko SH, Zimmet P, Son HY. Epidemic obesity and type 2 diabetes in Asia. Lancet. 2006 Nov 11;368(9548):1681-8. doi: 10.1016/S0140-6736(06)69703-1. PMID 17098087
- [Background] Villegas R, Shu XO, Gao YT, Yang G, Elasy T, Li H, Zheng W. Vegetable but not fruit consumption reduces the risk of type 2 diabetes in Chinese women. J Nutr. 2008 Mar;138(3):574-80. doi: 10.1093/jn/138.3.574. PMID 18287369
- [Background] Sargeant LA, Khaw KT, Bingham S, Day NE, Luben RN, Oakes S, Welch A, Wareham NJ. Fruit and vegetable intake and population glycosylated haemoglobin levels: the EPIC-Norfolk Study. Eur J Clin Nutr. 2001 May;55(5):342-8. doi: 10.1038/sj.ejcn.1601162. PMID 11378807
- [Background] Stratton IM, Adler AI, Neil HA, Matthews DR, Manley SE, Cull CA, Hadden D, Turner RC, Holman RR. Association of glycaemia with macrovascular and microvascular complications of type 2 diabetes (UKPDS 35): prospective observational study. BMJ. 2000 Aug 12;321(7258):405-12. doi: 10.1136/bmj.321.7258.405. PMID 10938048
- [Background] Riccardi G, Rivellese AA, Giacco R. Role of glycemic index and glycemic load in the healthy state, in prediabetes, and in diabetes. Am J Clin Nutr. 2008 Jan;87(1):269S-274S. doi: 10.1093/ajcn/87.1.269S. PMID 18175767
- [Background] Bell SJ, Sears B. Low-glycemic-load diets: impact on obesity and chronic diseases. Crit Rev Food Sci Nutr. 2003;43(4):357-77. doi: 10.1080/10408690390826554. PMID 12940416
- [Background] Liu S, Chou EL. Dietary glycemic load and type 2 diabetes: modeling the glucose-raising potential of carbohydrates for prevention. Am J Clin Nutr. 2010 Oct;92(4):675-7. doi: 10.3945/ajcn.2010.30187. Epub 2010 Sep 1. No abstract available. PMID 20810974
- [Background] Jimenez-Monreal AM, Garcia-Diz L, Martinez-Tome M, Mariscal M, Murcia MA. Influence of cooking methods on antioxidant activity of vegetables. J Food Sci. 2009 Apr;74(3):H97-H103. doi: 10.1111/j.1750-3841.2009.01091.x. PMID 19397724
- [Background] Salinero-Fort MA, Carrillo-de Santa Pau E, Arrieta-Blanco FJ, Abanades-Herranz JC, Martin-Madrazo C, Rodes-Soldevila B, de Burgos-Lunar C. Effectiveness of PRECEDE model for health education on changes and level of control of HbA1c, blood pressure, lipids, and body mass index in patients with type 2 diabetes mellitus. BMC Public Health. 2011 Apr 28;11:267. doi: 10.1186/1471-2458-11-267. PMID 21524316